CLINICAL TRIAL: NCT00481884
Title: Phase III Trial to Compare RadiaPlexRx Hydrogel and Standard-of-Care for Radiation Dermatitis in Breast Cancer Patients
Brief Title: Comparing RadiaPlexRx Hydrogel and Standard-of-Care for Radiation Dermatitis in Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-0827
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2012-01

CONDITIONS: Radiation Dermatitis
Keywords: Breast Cancer; Radiation Dermatitis; RadiaPlexRx Gel; Aquaphor
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RadiaPlexRx Gel (Experimental): RadiaPlexRx Gel for application to one half of irradiated breast skin, determined by a randomization process.
  Interventions: Other: RadiaPlexRx Gel
- Aquaphor Gel (Active Comparator): Aquaphor Gel for application to one half of irradiated breast skin, determined by a randomization process.
  Interventions: Other: Aquaphor Gel

INTERVENTIONS:
Other: RadiaPlexRx Gel — RadiaPlexRx Gel: The treated breast is divided into two vertical halves during the simulation using skin marker (medial and lateral halves). Patients are given detailed instructions to apply RadiaPlexRx gel topically 3 Times Daily to one half of the irradiated breast skin and the control, Aquaphor gel, to the other half of irradiated breast skin. This is determined through randomization process.
  Arms: RadiaPlexRx Gel
Other: Aquaphor Gel — Aquaphor Gel: The treated breast is divided into two vertical halves during the simulation using skin marker (medial and lateral halves). Patients are given detailed instructions to apply Aquaphor gel topically 3 Times Daily to one half of the irradiated breast skin and the experimental, RadiaPlexRx gel, to the other half of irradiated breast skin. This is determined through randomization process.
  Arms: Aquaphor Gel

SUMMARY:
Primary Objective:

To determine if RadiaPlexRx Hydrogel can reduce the development of grade 2 or higher radiation dermatitis in breast cancer from adjuvant radiation when compared to a petroleum-based gel (Aquaphor) commonly used as best supportive care.

DETAILED DESCRIPTION:
The Study Gels:

RadiaPlexRx (requires a prescription) and Aquaphor (over-the-counter) are both gels that are designed to treat irradiated (received radiation) breast skin.

These 2 gels contain different ingredients that may make one gel better than the other to treat irradiated breast skin. RadiaPlexRx contains hyaluronic acid (an ingredient found naturally in skin), aloe vera, and other ingredients that help the skin heal. Aquaphor is made of mostly petroleum that helps protect the skin.

Application of Study Gels:

If you decide to participate in this study, the following steps will be taken:

* You will be given detailed instructions on how to apply both of the gels. You should not apply other gels or lotions on the areas of skin where you will be instructed to apply the study gels, unless you are instructed to do so by the treating doctor.
* You will receive a supply of both gels (in tubes) with enough to last for the length of your treatment. You will know which gel is which, but each gel will be labeled with "outer" or "inner" so that you will know which gel to use on which side. You should not tell your treating doctor which side of the breast skin is being treated with which gel so that a fair comparison of the gels can be made.
* You will apply 1 gel to the outer side of the irradiated breast skin and the other gel to the inner side of the irradiated breast skin.
* If you experience any kind of allergic reaction (such as a rash) to the study gels, you should notify the study doctor or study staff immediately.

Schedule for Study Gels:

You will need to follow the schedule for applying the gels as follows:

* You will need to apply both gels starting 1 day before the start of radiation treatments.
* You will then need to apply both gels for 6 weeks during radiation treatment.
* During the study period (1 day before the start of radiation treatment, during 6 weeks of radiation treatment), you will need to apply both gels 3 times (in the morning, afternoon, and evening just before going to sleep) each day at home.
* During the days that you receive radiation treatment, you will be asked to apply the gels immediately after you receive your radiation treatment. This will count as 1 of the 3 daily gel applications.

Clinic Visits:

You will have the following tests done during your clinic visits:

* Three (3) sets of photos of your breast skin will be taken (before radiation starts and during Weeks 3 and 6 of radiation therapy treatment).
* During Weeks 1 through 6, you will go to the clinic to have your skin checked by your treating physician to learn the effects of each gel on your symptoms. .
* You will need to return any empty tubes of study gel so that new tubes can be given if you will need more.

Length of Study:

If the treating doctor sees that the irradiated breast skin reacts poorly (does not improve or gets worse) or you experience any intolerable side effects, you will be taken off this study. Otherwise, the total time on this study is about 6 weeks.

End-of-Study:

-During your last week of radiation therapy treatment you will be asked to fill out a questionnaire about how you felt about each gel.

This is an investigational study. RadiaPlexRx and Aquaphor are both FDA approved and commercially available. Up to 92 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically-confirmed carcinoma of breast (all subtypes are permitted)
2. Patient has breast conserving surgery (lumpectomy) for breast cancer with negative surgical margin
3. Stage Tis,0-3 N0-2 M0
4. Patient will receive irradiation of whole breast. An additional field to treat the supraclavicular / axillary apex lymphatics is allowed, but a separate field to treat the internal mammary chain nodes is not allowed
5. The breast will receive radiation dose greater than or equal to 50 Gy, with or without a boost field to give additional dose to the tumor bed
6. Patient wears bras with cup size larger than A
7. Patient signs informed consent

Exclusion Criteria:

1. Breast cancer treatment with mastectomy
2. Stage T4 breast cancer
3. Patient will require the use of tissue-equivalent bolus during radiation treatment or double treatment of junctions of radiation treatment fields
4. Patient will require treatment to the internal mammary chain lymph node bed using a separate radiation electron field
5. Patient is planned for partial-breast irradiation or Mammo-site treatment.
6. Patient has unhealed wound or rash in the radiation field
7. Patient has allergy to RadiaPlexRx or aloe vera
8. Patient has systemic lupus erythematosus or scleroderma that increases the risk of radiation dermatitis development
9. Patient will receive concurrent chemotherapy with radiation. (Patient is allowed to take concurrent hormonal therapy or Herceptin® [Trastuzumab])
10. Planned accelerated fractionation.
11. Planned radiation therapy to the bilateral breasts
12. Planned breast irradiation in the prone position

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients using RadiaPlexRx Hydrogel that developed grade 2 or higher radiation dermatitis in breast cancer from adjuvant radiation compared to a petroleum-based gel (Aquaphor) commonly used as best supportive care | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Buchholz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org